CLINICAL TRIAL: NCT05803837
Title: Effects of Concave Thoracoplasty on Chest Circumference and Ventilatory Function in Adolescence With Idiopathic Scoliosis
Brief Title: Thoracotomy Effects on Pulmonary Function Test and Chest Expansion
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Takey Ahmed, Asssociate Professor, Cairo University
Other Study IDs: Thoracotomy
Record Dates: First submitted 2023-02-07; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: lung functions and thoracotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention group: one group

SUMMARY:
The purpose of the present study was to investigate the effect that corrective surgery for scoliosis would have on pulmonary function as well as the circumference of the chest. As a result, the current investigation was carried out on thirty individuals who had idiopathic scoliosis and had been admitted to the hospital. Before the surgery, after it had been completed (on the fifth day), and again three months later, the pulmonary function was tested.

DETAILED DESCRIPTION:
The purpose of this study was to see how corrective scoliosis surgery affected pulmonary function and chest circumference. As a result, the current investigation was carried out on 30 individuals brought to the hospital with idiopathic scoliosis. The pulmonary function was assessed before surgery, on the fifth day following surgery, and three months thereafter.

ELIGIBILITY:
Inclusion Criteria:

• Adolescent idiopathic scoliosis

Exclusion Criteria:

* smoking.
* Associated comorbidity that affects PFT.
* Any contraindication interfering with performing spirometry.

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: thirty patients Participants have received a good explanation of the treatment and measurement device. aged between 12 and 18 years with AIS; the patients were admitted to hospital
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
chest expansion | 10 months
  chest circumference meaurement
PFT | 10 months for each parameter
  PULMONARY FUNCTION TEST
  * Vital capacity (Liter).
  * Forced VITAL Capacity (Liter).
  * Maximal voluntary breathing (Liter).

SECONDARY OUTCOMES:
cobb angle | 10 months
  In terms of measuring the major curve Cobb's angle, patient in a standing posterior-anterior (PA) radiograph, the angle is composed of two intersecting lines: the upper endplate of the main thoracic curve upper vertebra and the lower endplate of the main curve lower vertebra. These lines meet at the point where the upper endplate of the main thoracic curve upper vertebra and the lower endplate of the main curve lower vertebra meet.

CONTACTS AND LOCATIONS:
Overall Officials: nisreen moh elnahass, Prof, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rao KE, Krodel D, Toaz EE, Fanelli J, Hajduk J, Kato K, Rychlik K, King E, Sarwark J, Grayhack J, Burjek NE. Introduction of an enhanced recovery pathway results in decreased length of stay in patients with adolescent idiopathic scoliosis undergoing posterior spinal fusion: A description of implementation strategies and retrospective before-and-after study of outcomes. J Clin Anesth. 2021 Dec;75:110493. doi: 10.1016/j.jclinane.2021.110493. Epub 2021 Sep 2. PMID 34482261